CLINICAL TRIAL: NCT02103062
Title: A SINGLE ARM PHASE 2 STUDY TO EVALUATE THE SAFETY AND EFFICACY OF Nab®-PACLITAXEL, IN SUBJECTS WITH PREVIOUSLY TREATED METASTATIC COLORECTAL CANCER
Brief Title: Phase 2 Study With Abraxane (Nab®Paclitaxel) in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-COLO-001
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Neoplasms
Keywords: Metastatic Colorectal Cancer; nab®Paclitaxel; Response Evaluation in Solid Tumors; Progression Free Survival; Overall Survival; Duration of Response; RAS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abraxane (nab®paclitaxel) (Experimental): Abraxane (nab®paclitaxel) 125 milligrams per meter squared on days 1, 8 and 15 of a 28 day cycle
  Interventions: Drug: ABI-007

INTERVENTIONS:
Drug: ABI-007
  Other Names: Abraxane (nab®paclitaxel)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Abraxane (nab-paclitaxel) in subjects with previously treated metastatic colorectal cancer. Subjects will be placed into two separate cohorts based on their RAS mutation status.

DETAILED DESCRIPTION:
ABI-007-COLO-001 is a Phase 2, single arm, open label, multicenter study to evaluate the efficacy and safety of Abraxane (nab-paclitaxel) given on days 1, 8 and 15 of a 28 day cycle in subjects with previously treated metastatic colorectal cancer. Subjects will be enrolled into cohorts by RAS mutation status (wildtype or mutated). Stage 1 in a given cohort will enroll 15 subjects in the Intention to Treat population and if more than 8 subjects have Progression Free Survival at the 8 week assessment, then Stage 2 will open in the respective cohort. Stage 2 will enroll an additional 28 subjects for a total of 43 subjects in each cohort. The study will be positive if more than 26 subjects with Progression Free Survival at the 8 week assessment are observed in 43 subjects per cohort. Interim analysis after Stage 1 did not meet protocol defined criteria to proceed to Stage 2. Patients currently enrolled will be followed for Progression Free Survival and until 28 days after last dose, secondary endpoints including overall survival will not be followed

ELIGIBILITY:
Inclusion Criteria: - 1. Subject is ≥ 18 years old at the time of signing the Informed Consent Form 2. Subject has histological or cytological diagnosis of adenocarcinoma of the colon or rectum, with evidence of metastasis 3. Subject has a known KRAS mutation status (mutated or wild-type). NRAS mutation status may be unknown. 4. Subject has documented disease progression ≤ 2 months after the last administration of the last standard therapy. a. Subjects treated with oxaliplatin in the adjuvant setting, should have progressed during or within 6 months of completion of adjuvant therapy 5. Subject has either received prior treatment or was not a candidate for prior treatment, with fluoropyrimidine, oxaliplatin, irinotecan and an anti-VEGF therapy (e.g. bevacizumab or ziv-aflibercept); and if RAS wild-type tumors, an anti-EGFR therapy (e.g. cetuximab or panitumumab). 6. Subject has Eastern Cooperative Oncology Group performance status 0 or 1 7. Subject has radiographically-documented measurable disease, as per Response Evaluation Criteria in Solid Tumors version 1.1 criteria 8. Subject has adequate organ functions, evidenced by the following: a. Aspartate Aminotransferase (SGOT), Alanine Transaminase (SGPT) ≤ 2.5 × upper limit of normal range, or < 5 x upper limit of normal range if liver metastasis present b. Total bilirubin ≤ 1.5 × upper limit of normal range c. Creatinine ≤ 1.5 × upper limit of normal range 9. Subject has adequate bone marrow function, evidenced by the following: a. Absolute neutrophil count ≥ 1.5 × 109 cells/millimeters3 b. Platelets ≥ 100 × 109 cells/millimeters3 (transfusion independent, defined as not receiving platelet transfusions within 7 days prior to laboratory sample) c. Hemoglobin ≥ 9 grams/decilitre (transfusion is permitted to fulfill this criterion) 10. Females of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must: a. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting Investigational Product therapy (including dose interruptions), and for 3 months following the last dose of Investigational Product; and b. Have a negative serum pregnancy test (β -human Chorionic Gonadotrophin) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact. * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Note: Periodic abstinence (e.g, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. 11. Male subjects must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following Investigational Product discontinuation, even if he has undergone a successful vasectomy. 12. Subject must understand and voluntarily sign an Informed Consent Form prior to any study related assessments or procedures being conducted. 13. Subject must be able to adhere to the study visit schedule and other protocol requirements. Exclusion Criteria: - 1. Subject has current or a history of brain metastasis. In subjects who are symptomatic, a brain scan is required to exclude metastasis. 2. Subject has ≥ National Cancer Institute Common Terminology Criteria for Adverse Events grade 2 peripheral neuropathy at screening 3. Subject has had prior treatment with regorafenib 4. Subject has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting Investigational Product, and/or from whom ≥ 30% of the bone marrow was irradiated. Radiation therapy to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed. 5. Subject has had major surgery within 14 days prior to starting Investigational Product or has not recovered from postoperative complications 6. Subject has not recovered from the acute toxic effects of prior anticancer therapy, radiation or major /significant trauma 7. Subject has a history of allergy or hypersensitivity to nab-paclitaxel or any of the excipients 8. Subject has a known history of the following within 6 months prior to enrollment (the decision to include the subject in the study): a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or Electrocardiogram abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder 9. Subject has a known infection with hepatitis B or C, or history of human immunodeficiency virus infection, or subject receiving immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications 10. Subject has an active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment 11. Subject has any other malignancy within 5 years prior to enrolment, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, or non-melanomatous skin cancer (all treatment of which should have been completed 6 months prior to enrollment) 12. Subject has a history of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa) 13. Subject has a history of interstitial lung disease , history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies 14. Subject has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate subject participation in the clinical study (e.g. chronic pancreatitis, chronic active hepatitis, etc.) 15. Subject is enrolled in any other clinical protocol or investigational study with an interventional agent or assessments that may interfere with study procedures 16. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study 17. Subject has any condition that confounds the ability to interpret data from the study 18. Subject is unwilling or unable to comply with study procedures 19. Subject is a pregnant or nursing female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2014-11-10 (Actual); Study Completion 2015-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Romano, MD, Study Director — Celgene
Locations (6):
- France (6):
  - Centre Oscar Lambret, Dept. de Cancerologie Digestive et Urologique, Lille
  - Centre Regional de Lutte contre le Cancer Val d'Aurelle, Montpellier
  - Institut Curie, Saint-Cloud
  - CRLCC Centre Rene Gauducheau, Saint-Herblain
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy Hematologie, Villejuif

REFERENCES:
- [Derived] Ducreux M, Bennouna J, Adenis A, Conroy T, Lievre A, Portales F, Jeanes J, Li L, Romano A. Efficacy and safety of nab-paclitaxel in patients with previously treated metastatic colorectal cancer: a phase II COLO-001 trial. Cancer Chemother Pharmacol. 2017 Jan;79(1):9-16. doi: 10.1007/s00280-016-3193-5. Epub 2016 Nov 19. PMID 27866244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have been previously treated and must have had radiologically documented measurable disease, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and disease progression ≤ 2 months after the last delivery of the last standard therapy. They were enrolled by family of oncogenic proteins (RAS) mutation status .
Pre-assignment Details: An efficacy analysis was conducted based on the data available for those accrued in each of the cohorts enrolled (Stage 1) between May-September 2014. The data from the primary efficacy endpoint met the stopping criteria defined by the Simon 2-stage design, which did not support further assessment of nab-paclitaxel; the study was stopped early.
Groups:
- RAS Wildtype: Nab®-Paclitaxel; RAS Mutated: Nab®-Paclitaxel: nab®-paclitaxel 125 mg/m^2 on days 1, 8 and 15 of every 28 day cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel
Started | 18 | 23
Safety Population | 18 (Includes participants who received at least one dose of study drug.) | 23 (Includes participants who received at least one dose of study drug.)
Intent to Treat Population | 17 (Includes participants who met all eligibility criteria and received at least one dose of study drug.) | 20 (Includes participants who met all eligibility criteria and received at least one dose of study drug.)
Completed | 0 | 0
Not Completed | 18 | 23
Not completed — Adverse Event | 1 | 2
Not completed — Progressive Disease | 17 | 20
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Includes participants who met all eligibility criteria and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12.34) | 61.9 (10.56) | 63.0 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate as Measured at Week 8
Description: PFS rate was measured by Investigator Assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 from the start of study treatment to disease progression or death from any cause, whichever occurred first.
Time Frame: At week 8 assessment period; up to 56 days
Population: Per the Simon 2-stage design, only 30 participants from Stage 1 (the first 15 participants in the Intent to Treat (ITT) population from each cohort) were included. The ITT population was defined as those who received treatment and met all eligibility criteria; four ineligible participants were excluded based on the protocol deviations/violations
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel
Number analyzed (Participants) | 15 | 15
percentage of participants | 20 [4 to 48] | 20 [4 to 48]

2. Secondary Outcome: Percentage of Participants With Stable Disease for ≥ 8 Weeks, or Complete or Partial Response According to RECIST Version 1.1; Disease Control Rate (DCR)
Description: DCR was defined as the combined incidence of stable disease confirmed CR or PR and stable disease (SD) measured at the Week 8 assessment or later.
Time Frame: At week 8 and later; up to day 241
Population: ITT Population defined as participants who received treatment and met all eligibility criteria
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel
Number analyzed (Participants) | 17 | 20
Percentage of participants | 18 [4 to 43] | 15 [3 to 38]

3. Secondary Outcome: Overall Survival
Description: Overall Survival was the time from the first dose of study drug to patient death from any cause.
Time Frame: Up to 241 days
Population: The data from the primary efficacy endpoint met the stopping criteria defined by the Simon 2-stage design, which did not support further assessment of nab-paclitaxel as a monotherapy in the analysis of this group of participants. The study was stopped early and the analysis of overall survival was not performed.
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the combined incidence of Complete Response (CR) and Partial Response (PR), confirmed no less than 4 weeks after the criteria for response were first met based on RECIST 1.1. Tumor responses were assessed every 2 cycles using RECIST 1.1 and defined as: • Complete response-disappearance of all target lesions • Partial response- At least a 30% decrease in the sum of diameters of target lesions from baseline • Stable disease-neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for Progressive disease (PD) • Progressive Disease- At least a 20% increase in the sum of diameters of target lesions from nadir.
Time Frame: Up to 241 days
Population: ITT population defined as participants who received treatment and met all eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel
Number analyzed (Participants) | 17 | 20
percentage of participants | 0 [NA to NA] — NA because no participants experienced a CR or PR so the overall response rate in this study was zero. | 0 [NA to NA] — NA because no participants experienced a CR or PR so the overall response rate in this study was zero.

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the time from the first tumor assessment when the confirmed CR/PR response criterion was met to the date of disease progression based on investigational assessment following RECIST 1.1.
Time Frame: Up to 241 days
Population: The data from the primary efficacy endpoint met the stopping criteria defined by the Simon 2-stage design, which did not support further assessment of nab-paclitaxel as a monotherapy in the analysis of this group of participants. Duration of response was not analyzed as there were no responders observed in the study.
Groups:
- RAS Wildtype Abraxane (Nab®-Paclitaxel); RAS Mutated Abraxane (Nab®-Paclitaxel): Abraxane (nab®-paclitaxel) 125 mg/m^2 on days 1, 8 and 15 of every 28 day cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
Arm/Group | RAS Wildtype Abraxane (Nab®-Paclitaxel) | RAS Mutated Abraxane (Nab®-Paclitaxel)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Adverse Events
Description: A treatment emergent adverse events (TEAE) was defined as any AE occurring or worsening on or after the first dose of study drug and within 28 days after the last dose of study drug. A TESAE is defined as any serious adverse event (SAE) occurring or worsening on or after the first dose of study drug and within 28 days after the last dose of study drug. Safety and Severity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0; Severity of AEs were graded (including second primary malignancies) as Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Lifethreatening; Grade 5-Fatal;
Time Frame: Time of the first dose of study treatment to 28 days after the last dose of study drug; maximum treatment duration was 24 weeks
Population: Safety population includes all participants who received at least one dose of study treatment
Measure: Number; unit: participants
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel
Number analyzed (Participants) | 18 | 23
participants
  Any TEAE | 18 | 23
  ≥1 or more related TEAE | 17 | 21
  ≥1 TEAE with Grade 3-4 | 12 | 18
  ≥1 treatment related TEAE with Grade 3 or 4 | 9 | 12
  ≥1 or TEAE Grade 3 or higher | 12 | 18
  ≥1 treatment related TEAE with Grade 3 or higher | 9 | 12
  Any Serious TEAE | 5 | 10
  ≥1 or more related serious TEAE | 2 | 0
  ≥1TEAE with Action of Study Drug Withdrawn | 1 | 2
  ≥1treatment related TEAE WhereStudy Drug Withdrawn | 1 | 0
  ≥1TEAE with Action of Study Drug Reduced | 7 | 4
  ≥1 treatment related TEAE Where Study Drug Reduced | 6 | 4
  ≥1TEAE with study dose Interrupted | 7 | 8
  ≥1 treatment related TEAE w Study Drug Interrupted | 6 | 6
  ≥1TEAE with outcome of death | 0 | 1

7. Other Pre Specified Outcome: Kaplan Meier Estimate of PFS by Investigator Assessment
Description: PFS was measured as time from the date of first dose to the date of disease progression according to RECIST 1.1 or death from any cause, whichever was earlier.
Time Frame: Up to 241 days
Population: Intent-to-treat Population defined as participants who received treatment and met all eligibility criteria
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel
Number analyzed (Participants) | 17 | 20
weeks | 8.1 [7.71 to 8.57] | 7.9 [7.57 to 8.00]

ADVERSE EVENTS:
Time Frame: All adverse events were recorded and monitored by the investigator from the time the informed consent was signed to 28 days after the last dose of study treatment or the End of Treatment, whichever was later; maximum treatment duration was 24 weeks
Arm/Group | RAS Wildtype: Nab®-Paclitaxel | RAS Mutated: Nab®-Paclitaxel
Serious Adverse Events (participants affected / at risk) | 5/18 | 10/23
Other Adverse Events (participants affected / at risk) | 18/18 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAS Wildtype: Nab®-Paclitaxel (N=18) | RAS Mutated: Nab®-Paclitaxel (N=23)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Catheter site haematoma (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 2
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAS Wildtype: Nab®-Paclitaxel (N=18) | RAS Mutated: Nab®-Paclitaxel (N=23)
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2
Chapped lips (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 9
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 6 | 5
Vomiting (Gastrointestinal disorders) | 0 | 6
Asthenia (General disorders) | 16 | 17
Fatigue (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 6
Pyrexia (General disorders) | 3 | 4
Xerosis (General disorders) | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 3 | 3
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 2
Paronychia (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 4
Neuropathy peripheral (Nervous system disorders) | 4 | 4
Neurotoxicity (Nervous system disorders) | 2 | 1
Paraesthesia (Nervous system disorders) | 6 | 2
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 5
Sleep disorder (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 9
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 2 | 0
Lymphoedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally sixty (60) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.